CLINICAL TRIAL: NCT01968083
Title: A Phase I Study of the Safety and Immunogenicity of a Single Dose of the Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine RSV cps2, Lot RSV#005A, Delivered as Nose Drops to RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Evaluating the Safety and Immune Response to a Single Dose of a Respiratory Syncytial Virus (RSV) Vaccine in RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P1114; 11948 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2017-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSV cps2 Vaccine (Experimental): Participants will receive one dose of the RSV cps2 vaccine administered as nose drops at study entry.
  Interventions: Biological: RSV cps2 Vaccine
- Placebo (Placebo Comparator): Participants will receive one dose of placebo administered as nose drops at study entry.
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: RSV cps2 Vaccine — 10^5.3 plaque forming units (PFUs) or RSV cps2 vaccine will be administered as nose drops (0.25 mL per nostril, for a total of 0.5 mL).
  Arms: RSV cps2 Vaccine
Biological: Placebo Vaccine — Placebo vaccine will be administered as nose drops (0.25 mL per nostril, for a total of 0.5 mL).
  Arms: Placebo

SUMMARY:
Human respiratory syncytial virus (RSV) is a common cause of respiratory illness in infants and children. This study will evaluate the safety and immune response to an RSV vaccine in healthy RSV-naïve children.

DETAILED DESCRIPTION:
RSV is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age around the world. RSV illness can range from mild upper respiratory tract illness (URI) to severe LRI, including bronchiolitis and pneumonia. This study will evaluate the safety and immunogenicity of an RSV vaccine in healthy RSV-naïve children.

At study entry, participants will undergo a medical history review, physical examination, blood collection, and a nasal wash. Participants will be randomly assigned to receive the RSV vaccine or placebo at a 2:1 ratio, to be administered as nose drops. Participants will be actively monitored for 28 days following administration of vaccine or placebo; monitoring will include medical history reviews, clinical assessments, and at some visits, nasal washes. On the days when no study visit is scheduled, study researchers will contact participants' parents or guardians for medical follow-up. At a study visit on Day 56, participants will undergo a medical history review, blood collection, and a nasal wash procedure.

From November through March following each participant's study participation, parents or guardians will report respiratory and/or febrile illnesses on a weekly basis via telephone calls to study researchers. Participants may have additional study visits that may include blood collection and/or nasal wash procedures during this follow-up period.

This protocol is a companion study to CIR 285; a study being conducted by the Center for Immunization Research (CIR, Johns Hopkins, Baltimore), and the Laboratory of Infectious Diseases (NIAID, Bethesda). The protocols have identical primary and secondary objectives; immunization schedules; evaluation assays and schedules; safety monitoring and reporting. The protocols will vary slightly in site selection requirements, eligibility requirements and site monitoring. These are all operational issues modified to account for the IMPAACT sites' operations and infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians who demonstrate their understanding of the study (by taking a multiple choice questionnaire), sign the informed consent, and agree to vaccine administration following detailed explanation of the study
* Seronegative for RSV antibody, defined as a serum RSV neutralizing antibody titer less than 1:40 as determined within 42 days prior to enrollment/immunization
* Participant's history has been reviewed and participant has undergone a physical examination indicating that s/he is in good health
* In the view of the site investigator, the participant has received routine immunizations appropriate for their age
* Participant is expected to be available for the duration of the study
* For children born to HIV-infected women: two negative polymerase chain reaction (PCR) tests with one collected when greater than 1 month of age and one collected when greater than 4 months old, and no positive HIV PCR test; or two negative HIV antibody tests

Exclusion Criteria:

* Known or suspected impairment of immunological functions or HIV infection
* Receipt of immunosuppressive therapy including systemic corticosteroids within 30 days of study entry. NOTE: Topical steroids, topical antibiotic, and topical antifungal medications are acceptable within 24 hours of enrollment. May be reassessed after symptoms have resolved.
* Bone marrow/solid organ transplant recipients
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an RSV vaccine or previous receipt of or planned administration of any anti-RSV antibody product
* Previous serious vaccine-associated AE or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. Participants with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. Participants who had one episode of wheezing or received bronchodilator therapy for a single episode of illness in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may also be enrolled.
* Member of a household that includes an infant less than 6 months of age
* Member of a household that contains an immunocompromised individual (including, but not limited to: those with HIV-related immunodeficiency, defined as CD4 less than 300, or less than 15% if less than 5 years of age, measured within the previous 6 months; or any household members who have received chemotherapy within the last 12 months). Verbal report is sufficient documentation if the parent/guardian is confident of history.
* Attends day care with infants less than 6 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.
* Fever (rectal temperature of greater than or equal to 100.4°F [38°C]), or upper respiratory illness (rhinorrhea, cough, or pharyngitis) or nasal congestion significant enough to interfere with successful vaccination, or otitis media
* Participant has received any killed vaccine or live attenuated rotavirus vaccine within the last 2 weeks, any other live vaccine within the last 4 weeks, or gamma globulin (or other antibody products) within the past 3 months, or is scheduled to receive any immunization in the 28 days after enrollment
* Receipt of another investigational vaccine or investigational drug within 28 days of receiving this investigational RSV vaccine
* Participant has received antibiotics or systemic or nasal steroid therapy or other prescription medications for acute illness within 3 days of study entry. Permitted concomitant medications include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) topical steroids, topical antibiotics, and topical antifungal agents.
* Participant has received salicylate (aspirin) or salicylate-containing products within the past month
* Infants born at less than 37 weeks gestation and less than 1 year of age

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of vaccine-related solicited adverse events (AEs) that occur during the acute monitoring phase of the study (Days 0-28) | Measured through Day 28
  Frequency and severity of vaccine-related solicited adverse events (AEs) that occur during the acute monitoring phase of the study (Days 0-28)
Proportion of participants that develop 4-fold or greater rises in RSV neutralizing antibody titer following vaccination | Measured through study follow-up period, up to 1 year after study entry
  Antibody responses to the RSV F glycoprotein will also be assessed by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Coleen K. Cunningham, MD, Study Chair — Chief, Pediatric Infectious Diseases; T915, Children's Health Center
Locations (5):
- United States (5):
  - University of California, UC San Diego CRS, La Jolla, California
  - Miller Children's Hospital at Long Beach Memorial Medical Center, Long Beach, California
  - The Children's Hospital University of Colorado, Denver, Colorado
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois

REFERENCES:
- [Derived] Buchholz UJ, Cunningham CK, Muresan P, Gnanashanmugam D, Sato P, Siberry GK, Rexroad V, Valentine M, Perlowski C, Schappell E, Thumar B, Luongo C, Barr E, Aziz M, Yogev R, Spector SA, Collins PL, McFarland EJ, Karron RA; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) P1114 Study Team. Live Respiratory Syncytial Virus (RSV) Vaccine Candidate Containing Stabilized Temperature-Sensitivity Mutations Is Highly Attenuated in RSV-Seronegative Infants and Children. J Infect Dis. 2018 Apr 11;217(9):1338-1346. doi: 10.1093/infdis/jiy066. PMID 29509929